CLINICAL TRIAL: NCT04485767
Title: Preventing a Decline in Physical Function in Older Androgen-Deprived Men With Structured Exercise Training (RESIST-ADT Trial)
Brief Title: RESIST-ADT (Androgen Deprivation Therapy)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shehzad Basaria, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-193; R21AG065537 (NIH)
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer; Physical Function
Keywords: Prostate Cancer; Androgen Deprivation Therapy (ADT); Physical Function; Structured Exercise; Muscle Strength and Power
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pliability

STUDY DESIGN:
Intervention Model Description: Structured Resistance Exercise vs Control Exercise
Who Masked: Participant, Investigator
Masking Description: Participants, Investigators and Research Staff will remain blinded.
  Only exercise personnel and study statistician will be unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Resistance Training Exercise (Experimental): Men with prostate cancer who are about to begin androgen-deprivation therapy (ADT) will attend structured progressive resistance exercise training sessions 2 times/week for six months.
  Interventions: Behavioral: Progressive Resistance Training Exercise
- Flexibility and Balance Exercise (Active Comparator): Men with prostate cancer who are about to begin androgen-deprivation therapy (ADT) will attend flexibility and balance exercises training sessions 2 times/week for six months.
  Interventions: Behavioral: Flexibility and Balance Exercise

INTERVENTIONS:
Behavioral: Progressive Resistance Training Exercise — Progressive Resistance Training Exercise 2x weekly for 6 months.
  Arms: Progressive Resistance Training Exercise
Behavioral: Flexibility and Balance Exercise — Flexibility and Balance Exercise Training Exercise 2x weekly for 6 months.
  Arms: Flexibility and Balance Exercise

SUMMARY:
The overall goal of this study is to determine if implementing structured exercises prevent decline in muscle mass, muscle strength and physical function in men with prostate cancer undergoing androgen deprivation therapy (ADT). Our main hypothesis is that structured resistance exercise training in men undergoing ADT will preserve physical function assessed by loaded stair climbing power compared with the control group. The trial will also examine the efficacy of the exercise regimen on muscle strength, QOL and fatigue. The findings of this trial will lay the groundwork for definitive intervention trials to prevent frailty and falls in these men.

DETAILED DESCRIPTION:
This randomized, controlled, parallel group trial of 6-months duration is determining the efficacy of structured resistance exercise training in preventing the decline in physical function in older men with prostate cancer undergoing androgen deprivation therapy (ADT). It will compare the structured resistance exercise training with a control group of men undergoing flexibility and balance exercises training.

Men undergoing ADT for treatment of their prostate cancer experience a significant decline in muscle mass and muscle strength, which impacts their physical function. This predisposes them to frailty and a higher risk of falls. In addition to physical dysfunction, men undergoing ADT also experience a significant decrease in health-related quality of life and experience fatigue (tiredness).

This research study is taking a preventative approach to the physical function problems in men with prostate cancer by implementing exercise interventions before participants begin ADT that are specifically designed to improve muscle mass, muscle strength and physical function to lessen the impacts of muscle mass and strength decline.

The study includes a screening visit during which the following procedures will be conducted: Vitals, EKG, blood sample collection and a physical to determine eligibility. If qualified, participants will be randomly assigned to two different types of structured exercises: Resistance exercise training or flexibility and balance exercises. During the weekly exercise training 20 subjects will be assigned to the Exercise A group and 20 subjects to the Exercise B group. The exercise training sessions will occur approximately 2 times/week. In addition participants will also undergo DEXA scans, perform muscle strength testing and complete questionnaires at baseline, 3- and 6-month visits.

It is expected participants will be in this research study for up to 6 months. It is expected that about 40 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Men with active Prostate Cancer who are 60 years or older.
* Hormone-naive men about to undergo medical or surgical ADT.
* Planned ADT for at least 6 months.
* Life expectancy of at least 6 months from enrollment.
* Ability and willingness to provide informed consent.

Exclusion Criteria:

* Active medical conditions affecting participation in exercise training (limiting arthropathies, myopathies, severe peripheral vascular disease, or severe neuropathy).
* Cardiovascular disease (current angina, severe valvular disease, advanced congestive heart failure, arrhythmias, or stroke with residual muscular weakness).
* Prior hip or knee replacement.
* History of lower extremity fracture in the past 6 months.

Min Age: 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 21 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Loaded stair climb power | 6 months
  Compare the efficacy of a structured resistance exercise regimen vs a structured control regimen on loaded stair climb power. Assessment of physical function as measured by Loaded Stair Climbing Power.

SECONDARY OUTCOMES:
Body composition | 6 months
  Lean body mass measured by dual energy x-ray absorptiometry (DEXA)
Muscle strength and power | 6 months
  Maximal voluntary muscle strength in the lower extremities will be assessed by conducting the leg and chest press exercise by the 1-repetition maximum method and assessing loaded stair climb power.
Quality of Life (QOL) | 6 months
  Measured by SF-36 questionnaire a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being
Fatigue | 6 months
  Fatigue will be assessed by the Functional Assessment of Chronic Illness Therapy fatigue scale (FACIT-F).

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad Basaria, MD, Principal Investigator — Brigham and Women's Hospital; Thomas Storer, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Ernst M, Wagner C, Oeser A, Messer S, Wender A, Cryns N, Brockelmann PJ, Holtkamp U, Baumann FT, Wiskemann J, Monsef I, Scherer RW, Mishra SI, Skoetz N. Resistance training for fatigue in people with cancer. Cochrane Database Syst Rev. 2024 Nov 28;11(11):CD015518. doi: 10.1002/14651858.CD015518. PMID 39606939